CLINICAL TRIAL: NCT00513123
Title: A Pilot Study: Measurement of Digital Colposcopy for Fluorescence Spectroscopy of Cervical Intraepithelial Neoplasia
Brief Title: Measurement of Digital Colposcopy for Fluorescence Spectroscopy of Cervical Intraepithelial Neoplasia
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: GYN98-258
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Cervical Cancer
Keywords: Digital Colposcopy for Fluorescence; DCF; Fluorescence Spectroscopy; Digital Colposcopy; DC; Cervical Intraepithelial Neoplasia; Cervical Cancer; Cervix; Vagina; Lesions of the cervix; Precancerous lesions
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia | interventions — Colposcopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Digital Colposcopy: Digital Colposcopy for Fluorescence (DCF)
  Interventions: Procedure: Colposcopy

INTERVENTIONS:
Procedure: Colposcopy — As part of routine colposcopic evaluation, patients will undergo routine colposcopy with the digital colposcope (DC) will then be used to take an image of the vagina and cervix.

SUMMARY:
The overall objective of this study is to identify potential improvements for a noninvasive method of diagnosing dysplasia and neoplasia in the cervix using digital colposcopy for colposcopy for fluorescence spectroscopy.

Other Objectives:

* To measure digital fluorescence and reflectance images in vivo of sites in the human cervix.
* To evaluate the effect of acetic acid in the image contrast obtained.
* Compare the device performance to colposcopy and pathologic analysis of tissue removed at colposcopy.

DETAILED DESCRIPTION:
DCF may provide a better way to detect or treat lesions of the cervix. Women in the study will already be scheduled for colposcopy to detect or treat lesions of the cervix. (A colposcopy is an exam of the vagina and cervix using a magnifying lens).

DCF will be done during the routine colposcopy in the outpatient clinic. A digital colposcope (DC) device will be used to take a sequence of images of the cervix and vagina. (A DC is a digital camera connected to the colposcope with a specialized light source. It will shine light on the cervix and acquire a sequence images). The images will tell doctors about the cells and structure of the tissue. After the first set of images, acetic acid will be applied to the cervix so that lesions show up better, and 1-2 minutes later more readings will be taken.

Small samples of areas of abnormal tissue will be removed during colposcopy. Taking these tissue samples is a routine part of this type of exam. If patients are having colposcopy and loop electrosurgical excision procedure (LEEP treatment, one sample of normal tissue will be taken. (The cervix will be numbed for this procedure.) DCF images will be compared with lab findings from these samples. Before DCF is done, as standard of care, patients will have a complete history and physical exam, urine pregnancy test, pap smear, and cultures for gonorrhea, chlamydia and viral testing.

This is an investigational study. About 114 women will take part in this study. About 22 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 and older with an abnormal Pap

Exclusion Criteria:

* Pregnant individuals will be excluded from this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women 18 and older with an abnormal PAP.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2002-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
To study whether digital colposcopy for fluorescence (DCF) can perform better than standard methods to detect cancer of the cervix or precancerous lesions. | 7 Years

CONTACTS AND LOCATIONS:
Overall Officials: Michele Follen, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (5):
- United States (3):
  - Lyndon B. Johnson Hospital, Houston, Texas
  - U.T. Health Science Center, Houston, Texas
  - U.T.M.D. Anderson Cancer Center, Houston, Texas
- British Columbia Cancer Research Center, Vancouver, British Columbia, Canada
- University College Hospital, Ibadan, Oyo State, Nigeria

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org